CLINICAL TRIAL: NCT01498861
Title: A Double-Blind Study to Evaluate the Pharmacokinetics of an Oral Contraceptive Containing Norgestimate and Ethinyl Estradiol When Co-administered With Dolutegravir in Healthy Adult Female Subjects
Brief Title: Drug Interaction Study Between Dolutegravir and an Oral Contraceptive Containing Norgestimate and Ethinylestradiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 111855
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-04

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Moxifloxacin; dolutegravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Run-In Period (Other): Ortho-Cyclen for 21 days. Only for subjects who are not already taking Ortho-Cyclen prior to the study
  Interventions: Drug: Ortho-Cyclen
- Sequence AB (Experimental): Subjects will take Ortho-Cyclen once a day from Day 1-21 of their menstrual cycle. In addition they will take dolutegravir 50 mg twice a day from Days 1-10 and placebo twice a day from Day 12-21
  Interventions: Drug: Ortho-Cyclen; Drug: Dolutegravir; Drug: Placebo
- Sequence BA (Experimental): Subjects will take Ortho-Cyclen once a day from Day 1-21 of their menstrual cycle. In addition they will take placebo twice a day from Days 1-10 and dolutegravir 50 mg twice a day from Day 12-21
  Interventions: Drug: Ortho-Cyclen; Drug: Dolutegravir; Drug: Placebo

INTERVENTIONS:
Drug: Ortho-Cyclen — Ortho-cyclen is an oral contraceptive.
Drug: Dolutegravir — Dolutegravir is an experimental HIV drug
  Other Names: GSK1349572
  Arms: Sequence AB; Sequence BA
Drug: Placebo — Placebo is a tablet with no drug in it
  Arms: Sequence AB; Sequence BA

SUMMARY:
Dolutegravir (DTG, GSK1349572 is an integrase inhibitor that is currently in Phase 3 clinical development for the treatment of HIV infection. DTG will likely be used in women on oral contraceptives (OC) for birth control. Based on accumulated non-clinical and clinical drug metabolism and pharmacokinetic data, there is a low likelihood of drug interaction between DTG and most widely used OC drugs. The primary objective of this study is to evaluate the effect of DTG administration on the pharmacokinetics and pharmacodynamics of a commonly used oral contraceptive product, Ortho-Cyclen (combination of norgestimate and ethinyl estradiol), in healthy female subjects. Each subject will participate in a Run-in period (if needed), followed by two treatment periods. Approximately 16 subjects will be randomized in a cross-over fashion to either Ortho-Cyclen with DTG or Ortho-Cyclen with Placebo for 10 days and switch to the alternate treatment for another 10 days. Subjects will return to the study center for final follow up evaluations 7 - 14 days after the final dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin greater than or equal to 1.5 times the upper limit of normal (ULN)
* Healthy female subjects, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied except for ALT, alkaline phosphatase and bilirubin as above may be included only if the Investigator feels that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Female, between 18 and 40 years of age inclusive, at the time of signing the informed consent.
* Women of childbearing potential must use OC Ortho-Cyclen in combination with one of the following appropriate contraceptive methods:a)Complete abstinence from intercourse for at least 14 days prior to the first dose of investigational product (Day 1 of Period 1), throughout the study, and for the subsequent poststudy monitoring or; b) A barrier method plus a spermicide (e.g., condom or diaphragm with spermicidal foam/gel/cream/ suppository for at least 14 days prior to the first dose of investigational product [Day 1 of Period 1]) throughout the study, and for the subsequent poststudy monitoring or; c)Sterilization (vasectomy) of male partner prior to commencement of female subject's last normal menstrual period prior to administration of study drug, and the male partner is the sole partner for that female subject.
* The subject's BMI is 19 to 30 kg/m2 and body weight ≥50 kg (110 lbs) and <114 kg (<250 lbs);
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
* Single QTcB < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception (see inclusion criteria) from at least 14 days prior to the first dose of investigational product until completion of the follow-up visit;
* Pregnant females as determined by positive hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of any condition that would contraindicate OC administration (including hypertension, stroke, ischemic heart disease, venous thromboembolism or family history of thromboembolism, known factor V Leiden mutation or other gene mutations associated with increased risk of thromboembolism, migraine headaches, carcinoma of the breast, liver or endometrium, gallbladder disease, history of undiagnosed abnormal uterine bleeding, etc.).
* If heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Unwilling to abstain from tobacco use from the screening visit until the follow-up visit.
* Females with conditions or concurrent medications that could adversely affect hormone levels e.g. oopherectomies and females receiving drug eluting IUDs (e.g. Mirena).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
AUC(0-tau) of norelgestromin and ethinylestradiol after Ortho-Cyclen alone and after Ortho-Cyclen with dolutegravir | Up to 24 hours post-dose
  Samples will be collected at predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose on Days 10 and 21

SECONDARY OUTCOMES:
Safety and tolerability of all treatments as assessed by vital signs, AEs, and clinical laboratory tests | Up to 8 weeks
Composite of norelgestromin pharmacokinetic parameters on Day 10 and Day 21: Cmax, Cmin, tmax, tmin and half life | Up to 24 hours post dose
  Samples will be collected at predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, and 24 hours postdose on Days 10 and 21
Predose serum levels of luteinizing hormone and follicle stimulating hormone from Periods 1 and 2 | predose on Days 1, 10, 11, 21 and 22
  Samples will be collected at predose on Days 1, 10, 11, 21 and 22
Predose serum levels of progesterone from Periods 1 and 2 | predose on Days 1, 10, 11, 21 and 22
  Samples will be collected at predose on Days 1, 10, 11, 21 and 22
Composite of dolutegravir pharmacokinetic parameters on Day 10 and Day 21: AUC(0-t), Cmax, tmax, Cmin, C0, Ct and CL/F | Up to 12 hours post dose
  Samples will be collected at predose and at 1, 2, 3, 4, 6, 8, and 12 hours post dose on Day 10 and Day 21

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Miami, Florida, United States